CLINICAL TRIAL: NCT03425162
Title: Ultrasound Guided Anterior Quadratus Lumborum Block for Postoperative Pain After Percutaneous Nephrolithotomy: Randomized Controlled Trial
Brief Title: Ultrasound Guided Anterior Quadratus Lumborum Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BYIEAH
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Postoperative Pain; Ultrasound
Keywords: quadratus lumborum block; pain; ultrasound; percutaneous nephrolithotomy
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Morphine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: prospective,randomized,single blind
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A:Ultrasound guided unilateral anterior Quadratus Lumborum block with 20 ml %0.25 bupivacaine+PCA (morphine)
  Interventions: Drug: Morphine Sulfate; Procedure: Group A
- Group P (Sham Comparator): Group P:PCA (morphine)
  Interventions: Drug: Morphine Sulfate; Procedure: Group P

INTERVENTIONS:
Drug: Morphine Sulfate — patient-controlled analgesia (PCA) morphine
  Other Names: Morphine
Procedure: Group P — Group P:patient-controlled analgesia (PCA) morphine
  Arms: Group P
Procedure: Group A — Group A:Ultrasound guided unilateral anterior Quadratus Lumborum block with 20 ml %0.25 Bupivacaine
  Other Names: Bupivacaine
  Arms: Group A

SUMMARY:
Percutaneous nephrolithotomy (PNL) is frequently used today for renal stones. percutaneous nephrolithotomy (PNL) procedure has become the treatment of choice for many patients with symptomatic renal stones . Patients undergoing PNL suffer from acute postoperative pain, despite a multimodal analgesic regime.

This is a randomised controlled trial efficacy of the anterior Quadratus Lumborum Block (QLB) in terms of analgesic efficacy in patients who undergo percutaneous nephrolithotomy.

DETAILED DESCRIPTION:
Many analgesic procedures such as NSAID, opioid and regional anesthesia procedures are used as a part of multimodal analgesia for postoperative Percutaneous nephrolithotomy pain.

In this study we will use the ultrasound -guided anterior Quadratus Lumborum Block . Local anesthesic will be injected between quadratus lumborum muscle and psoas muscle with ultrasound.Analgesic effect of this block will be detected by using morphine consumption and visual analogue scale .

ELIGIBILITY:
Inclusion Criteria:

* Patients who were in the American Society of Anesthesiologists (ASA) I-III class and underwent elective Percutaneous nephrolithotomy

Exclusion Criteria:

* Previous history of opioid use preoperatively,

  * Allergy to local anesthetics,
  * The presence of any systemic infection,

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-08-18 (Actual); Study Completion 2018-08-18 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Postoperative 24 hours
  Visual Analog Scale was used for pain.Pain intensity was measured using 0-10 cm visual analogue scale (VAS). (0= no pain, 10=intolerable pain)

SECONDARY OUTCOMES:
morphine consumption | Postoperative 24 hours
  morphine consumption
side effect profile | Postoperative 24 hours
  side effect profile (Nausea and vomiting scale,Hypotension,Ramsay Sedation Scale)
  1. Nausea and vomiting scale (nausea-vomiting scale (NVS): 1. No nausea is present, 2. Mild nausea is present. 3. Severe nausea is present. 4. Vomiting is present) In case of a NVS score of >3, an anti-emetic drug was administered.
  2. Hypotension
  3. Ramsay Sedation Scale (Ramsay Sedation Scale (RSS) : 1. Anxiety, agitation are present; 2. Cooperated, awake; 3. Sedatized, response to commands; 4. Sleepy, immediately awoken by auditory stimulus or glabella tap; 5. Sleepy, deep response to auditory stimulus or glabella tap and 6. Sleepy, no response to auditory stimulus or glabella tap )
additional analgesic use | Postoperative 24 hours
  additional analgesic use

CONTACTS AND LOCATIONS:
Overall Officials: Korgün Ökmen, M.D, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- University of Health Sciences, Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Turkey (Türkiye)